CLINICAL TRIAL: NCT06953479
Title: MINMON-J: An Effectiveness Implementation Pilot Study Evaluating a Low-barrier Hepatitis C Treatment Model in a Jail Setting
Brief Title: Implementing Low-Barrier HCV Treatment in a Jail Setting
Acronym: MINMON-J
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Lifespan (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Justin Berk, Assistant Professor, Lifespan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 2240400; R34DA061732 (NIH)
Record Dates: First submitted 2025-04-16; First posted 2025-05-01 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: HEPATITIS C (HCV); Incarceration; Injection Drug Use; Implementation Science
Keywords: hepatitis c; incarceration; jail; injection drug use; minimal monitoring; MINMON; implementation science
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir; velpatasvir; sofosbuvir-velpatasvir drug combination; Community Health Workers

STUDY DESIGN:
Intervention Model Description: Pilot Single-Arm Hybrid Implementation-Effectiveness Study; adaptation of "Minimal Monitoring" HCV treatment model
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- MINMON-J (Experimental): Individuals in this arm will be provided the full-course treatment of sofosbuvir / velpatasvir for treatment of hepatitis C virus. They will also receive support from a Community Health Worker (CHW) to assist with community re-entry, medication adherence, and lab follow-up.
  Interventions: Drug: Sofosbuvir / Velpatasvir Oral Tablet [Epclusa]; Other: Community Health Worker

INTERVENTIONS:
Drug: Sofosbuvir / Velpatasvir Oral Tablet [Epclusa] — Individuals will receive a full course (i.e., 84 tablets) of Sofosbuvir / Velpatasvir 400/100mg tablets.
Other: Community Health Worker — Participants will receive support from a Community Health Worker which may include assistance with basic needs (transportation, housing, employment, vital documents, insurance re-activation) as well as medication adherence, patient navigation, and peer recovery support.
  Other Names: CHW

SUMMARY:
The goal of this clinical trial is to learn whether a low-barrier treatment program can help people with hepatitis C virus (HCV) who are in jail start and complete treatment more easily. This study focuses on adults at the Rhode Island Department of Corrections who have active HCV and are awaiting trial.

The study asks:

* Can a simplified, low-barrier HCV treatment program work in a jail setting?
* Do participants finish treatment and get cured using this approach?

All participants will receive a 12-week course of the HCV medication sofosbuvir/velpatasvir (Epclusa). If they are released before completing treatment, they will take the remaining doses with them. Community Health Workers (CHWs) will help support participants after release, including reminding them to take medications and helping them get follow-up lab work.

Researchers will measure:

* Whether participants are cured of HCV
* Whether the treatment approach is easy to use (feasible), acceptable, and followed correctly (fidelity)
* Whether the program could be used in other jails or expanded in the future

This study may help bring HCV treatment to more people in jail, reduce community spread of the virus, and support national goals to eliminate HCV.

DETAILED DESCRIPTION:
This is a hybrid effectiveness-implementation pilot study testing a simplified model of hepatitis C virus (HCV) treatment called MINMON-J, based on the successful "minimal monitoring" approach used in community settings. The study takes place at the Rhode Island Department of Corrections (RIDOC), a statewide unified jail and prison system. The goal is to assess whether low-barrier HCV treatment can be feasible, acceptable, and effective when started in jail, especially for individuals who inject drugs.

Participants will receive a full 12-week course of sofosbuvir/velpatasvir (Epclusa) with no lab monitoring required during treatment. Those released before completing treatment will be given take-home medication and supported by Community Health Workers (CHWs) post-release. CHWs will check in with participants, support medication adherence, and help coordinate follow-up testing.

The study will enroll 40 adults with active HCV who are awaiting trial and meet other medical and safety criteria. Implementation outcomes will be assessed using the PRISM/RE-AIM framework. These include:

Feasibility: Can the treatment be delivered as planned in the jail setting? Acceptability: Do participants and providers find the program acceptable? Fidelity: Do participants take the medication as prescribed? Effectiveness: Are participants cured of HCV (measured by SVR12)? Maintenance: Do participants remain engaged in care or avoid reinfection 6 months later?

Additional data will include participant demographics, adherence rates, and program costs (via the COINS framework). Participants and staff will also take part in qualitative interviews to understand their experience and identify ways to improve implementation. Results will inform a future larger trial and contribute to efforts to scale up HCV treatment in carceral settings as part of national HCV elimination efforts.

ELIGIBILITY:
Inclusion Criteria:

* Incarcerated individual at RIDOC
* Age ≥ 18 years
* Awaiting trial (i.e., not sentenced)
* English speaking
* Diagnosis of active HCV (HCV RNA >1000 IU/mL within 90 days prior to study entry)
* Treatment-naïve for current HCV infection
* No cirrhosis (FIB-4 Score <3.25 within 90 days prior to study entry)
* Self-report of injection drug use
* Ability and willingness to be contacted after jail release
* Verbal commitment to continue medication after discharge
* Desire to receive Sofosbuvir/Velpatasvir (Epclusa)

Exclusion Criteria:

* Cirrhosis (FIB-4 Score >3.25 within 90 days prior to study entry and/or clinical signs of cirrhosis)
* Positive for Hepatitis B surface antigen
* Actively pregnant or breastfeeding
* Known allergy/sensitivity to study drug components
* Acute or serious illness requiring hospitalization at enrollment
* Documented severe persistent mental illness (SPMI) by RIDOC
* Any clinical history of hepatic decompensation (e.g., ascites, SBP, HE, HRS, variceal bleeding)
* HIV-positive with active or acute AIDS-defining opportunistic infection within 90 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
HCV Cure Rate | Between 12 and 24 weeks after completion of HCV treatment
  HCV Cure Rate will be defined as achieving a Sustained Virological Response at 12 weeks after treatment completion (SVR12), assessed by an undetectable HCV RNA viral load measured via standard laboratory assay. An undetectable result indicates that the virus is no longer present in the blood and is considered the clinical definition of virologic cure.

SECONDARY OUTCOMES:
Implementation: Feasibility of Implementation Measure | Between 4 to 12 weeks post-implementation
  The Feasibility of Implementation Measure (FIM) is a validated 4-item Likert-scale tool assessing provider perceptions of the feasibility of implementing a specific intervention. Each item is scored from 1 (completely disagree) to 5 (completely agree), with higher scores indicating greater perceived feasibility. The total score ranges from 4 to 20. Mean FIM scores will be reported across participants. This will be administered to participating stakeholders.
Fidelity: In-facility Treatment Adherence | From enrollment to the end of treatment at 12 weeks
  Fidelity will be assessed by calculating the percentage of prescribed doses taken during the treatment period, based on in-facility medication dispensation data from the Rhode Island Department of Corrections (RIDOC) electronic medical record (EMR), Adherence will be reported both as a continuous variable (% of doses taken) and as a binary indicator (≥80% of prescribed daily doses taken during treatment). Missing doses will be quantified to assess treatment fidelity across care settings.
Fidelity: Community Treatment Adherence | From enrollment to the end of treatment at 12 weeks
  Fidelity will be assessed by calculating the percentage of prescribed doses taken during the treatment period, based on community adherence data collected by community health workers (CHWs) using the Brief Adherence Rating Scale (BARS). Adherence will be reported both as a continuous variable (% of doses taken) and as a binary indicator (≥80% of prescribed daily doses taken during treatment). Missing doses will be quantified to assess treatment fidelity across care settings.
Implementation: Acceptability of Implementation Measure | Between 4 to 12 weeks post-implementation
  Acceptability will be assessed using the validated 4-item Acceptability of Intervention Measure (AIM), which evaluates provider perceptions of how acceptable the intervention is. Each item is rated on a 5-point Likert scale ranging from 1 (completely disagree) to 5 (completely agree). Total scores range from 4 to 20, with higher scores indicating greater acceptability.

CONTACTS AND LOCATIONS:
Locations (1):
- Rhode Island Department of Corrections, Cranston, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Berk J, Fu ES, Murphy M, Akiyama MJ, Sulkowski M, Rich JD, Frank HE. MINMON-J: a hybrid implementation pilot study evaluating a low-barrier hepatitis C treatment model in a jail setting. BMJ Open. 2025 Sep 30;15(9):e104839. doi: 10.1136/bmjopen-2025-104839. PMID 41027703